CLINICAL TRIAL: NCT06852521
Title: Probing the Role of Feature Dimension Maps in Visual Cognition: Expt 3.1 (Pilot)
Brief Title: Probing the Role of Feature Dimension Maps in Visual Cognition: Manipulations of Relevant Locations on Salience Processing? (Expt 3.1 Pilot)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Santa Barbara (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-25-0048: 3.1 (Pilot); R01EY035300 (NIH)
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Basic Science: Visual Attention in Healthy Participants; Attention

STUDY DESIGN:
Intervention Model Description: This is a basic science study in which all participants will participate in all task conditions within each experiment (repeated-measures design).
Masking Description: Participants will typically be unaware of the conditions presented, though because these involve manipulations of stimuli or task demands, they may be aware of the manipulation. This is not expected to impact the primary outcome measures (e.g., behavioral performance).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manipulations of Relevant Locations (Expt 3.1 Pilot) (Experimental): Participants will complete a visual search task in which they will covertly search for a unique target item based on a specific feature dimension indicated at the start of the experiment (unique color, unique motion direction, unique shape) in an 8 item array. At the beginning of each trial, participants will be visually cued (e.g., an arrowhead around fixation) to the side of the display the target item will appear (left, right, up, down). A proportion of all trials will contain a task-irrelevant, singleton distractor defined in a non-target dimension (e.g., color target and motion distractor)
  Interventions: Other: Stimulus Properties: Target Location; Other: Stimulus Properties: Distractor Presence; Other: Stimulus properties: Cue Validity

INTERVENTIONS:
Other: Stimulus Properties: Target Location — The location of the target item in the display will be varied across trials (appear left, right, up, or down)
Other: Stimulus Properties: Distractor Presence — A proportion of all trials will contain a task-irrelevant, singleton distractor defined in a non-target dimension (e.g., color target and motion distractor)
Other: Stimulus properties: Cue Validity — Varied across trials, the validity of the cue will be determined by the match or mismatch between direction of the visual cue (an arrowhead around the fixation pointing to the right, left, up, or down) and actual target location

SUMMARY:
How do we know what's important to look at in the environment? Sometimes, we need to look at objects because they are 'salient' (for example, bright flashing lights of a police car, or the stripes of a venomous animal), while other times, we need to ignore irrelevant salient locations and focus only on locations we know to be 'relevant'. These behaviors are often explained by the use of 'priority maps' which index the relative importance of different locations in the visual environment based on both their salience and relevance. In this research, we aim to understand how these factors interact when determining what's important to look at. Specifically, we are evaluating the extent to which the visual system considers locations that are known to be irrelevant when considering the salience of objects. We're testing the hypothesis that the visual system always computes maps of salient locations within 'feature maps', but that activity from these maps is not read out to guide behavior for task-irrelevant locations. We'll have people look at displays containing colored shapes and/or moving dots and report aspects of the visual stimulus (e.g., orientation of a line within a particular stimulus). We'll measure response times across conditions in which we manipulate the presence/absence of salient distracting stimuli and provide various kinds of cues about the potential relevance of different locations on the screen.

The rationale is that by measuring changes in visual search behavior (and thus inferring computations performed on brain representations), we will determine how these aspects of simplified visual environments impact the brain's representation of important object locations. This will support future studies using brain imaging techniques aimed at identifying the neural mechanisms supporting the extraction of salient and relevant locations from visual scenes, which can inform future diagnosis/treatment of disorders which can impact our ability to perform visual search (e.g., schizophrenia, Alzheimer's disease).

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 55 years of age
* normal or corrected-to-normal vision

Exclusion Criteria:

• N/A

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Behavioral response (button press) | Through study completion, an average of two weeks
  Participants will be required to report the orientation of a line (horizontal or vertical) within the target via a speeded button press. The specific values of color, shape, and motion will vary randomly from trial to trial. Participants will complete separate sessions with each session directing participants to search for a different target feature dimension.
Gaze position | Through study completion, an average of two weeks
  The investigators will use the measured gaze position in (x,y) coordinates to verify stable fixation throughout the experiment. The data will be used to establish gaze fixation and/or track where participants look as they perform the visual search task. Trials with poor fixation performance may be excluded from further analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy C Sprague, Principal Investigator — University of California, Santa Barbara
Locations (1):
- University of California, Santa Barbara, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw behavioral data will be shared with researchers immediately upon publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available indefinitely beginning with publication of results
Access Criteria: Raw behavioral/eyetracking data will be publicly available on the lab's Open Science Framework page (https://osf.io/ufjzl/), and analysis code will be available on GitHub (an online tool for storing and managing code; github.com/SpragueLab)
URL: https://osf.io/ufjzl/

REFERENCES:
- [Background] Mackey WE, Winawer J, Curtis CE. Visual field map clusters in human frontoparietal cortex. Elife. 2017 Jun 19;6:e22974. doi: 10.7554/eLife.22974. PMID 28628004
- [Background] Hallenbeck GE, Sprague TC, Rahmati M, Sreenivasan KK, Curtis CE. Working memory representations in visual cortex mediate distraction effects. Nat Commun. 2021 Aug 5;12(1):4714. doi: 10.1038/s41467-021-24973-1. PMID 34354071
- [Background] Sprague TC, Itthipuripat S, Vo VA, Serences JT. Dissociable signatures of visual salience and behavioral relevance across attentional priority maps in human cortex. J Neurophysiol. 2018 Jun 1;119(6):2153-2165. doi: 10.1152/jn.00059.2018. Epub 2018 Feb 28. PMID 29488841
- [Background] Sprague TC, Adam KCS, Foster JJ, Rahmati M, Sutterer DW, Vo VA. Inverted Encoding Models Assay Population-Level Stimulus Representations, Not Single-Unit Neural Tuning. eNeuro. 2018 Jun 5;5(3):ENEURO.0098-18.2018. doi: 10.1523/ENEURO.0098-18.2018. eCollection 2018 May-Jun. No abstract available. PMID 29876523
- [Background] Sprague TC, Boynton GM, Serences JT. The Importance of Considering Model Choices When Interpreting Results in Computational Neuroimaging. eNeuro. 2019 Dec 20;6(6):ENEURO.0196-19.2019. doi: 10.1523/ENEURO.0196-19.2019. Print 2019 Nov/Dec. PMID 31772033
- [Background] Laumann TO, Gordon EM, Adeyemo B, Snyder AZ, Joo SJ, Chen MY, Gilmore AW, McDermott KB, Nelson SM, Dosenbach NU, Schlaggar BL, Mumford JA, Poldrack RA, Petersen SE. Functional System and Areal Organization of a Highly Sampled Individual Human Brain. Neuron. 2015 Aug 5;87(3):657-70. doi: 10.1016/j.neuron.2015.06.037. Epub 2015 Jul 23. PMID 26212711
- [Background] Allen EJ, St-Yves G, Wu Y, Breedlove JL, Prince JS, Dowdle LT, Nau M, Caron B, Pestilli F, Charest I, Hutchinson JB, Naselaris T, Kay K. A massive 7T fMRI dataset to bridge cognitive neuroscience and artificial intelligence. Nat Neurosci. 2022 Jan;25(1):116-126. doi: 10.1038/s41593-021-00962-x. Epub 2021 Dec 16. PMID 34916659
- [Background] Fedorenko E. The early origins and the growing popularity of the individualsubject analytic approach in human neuroscience. Current Opinion in Behavioral Sciences. 2021; 40:105-112.
- [Background] Naselaris T, Allen E, Kay K. Extensive sampling for complete models of individual brains. Current Opinion in Behavioral Sciences. 2021; 40:45-51.
- [Background] Poldrack RA. Diving into the deep end: a personal reflection on the MyConnectome study. Current Opinion in Behavioral Sciences. 2021; 40:1-4.
- [Background] Pritschet L, Taylor CM, Santander T, Jacobs EG. Applying dense-sampling methods to reveal dynamic endocrine modulation of the nervous system. Curr Opin Behav Sci. 2021 Aug;40:72-78. doi: 10.1016/j.cobeha.2021.01.012. Epub 2021 Feb 25. PMID 35369044
- [Background] Gratton C, Nelson SM, Gordon EM. Brain-behavior correlations: Two paths toward reliability. Neuron. 2022 May 4;110(9):1446-1449. doi: 10.1016/j.neuron.2022.04.018. PMID 35512638
- [Background] Smith PL, Little DR. Small is beautiful: In defense of the small-N design. Psychon Bull Rev. 2018 Dec;25(6):2083-2101. doi: 10.3758/s13423-018-1451-8. PMID 29557067
- [Background] Sprague TC, Serences JT. Attention modulates spatial priority maps in the human occipital, parietal and frontal cortices. Nat Neurosci. 2013 Dec;16(12):1879-87. doi: 10.1038/nn.3574. Epub 2013 Nov 10. PMID 24212672
- [Background] Itthipuripat S, Vo VA, Sprague TC, Serences JT. Value-driven attentional capture enhances distractor representations in early visual cortex. PLoS Biol. 2019 Aug 9;17(8):e3000186. doi: 10.1371/journal.pbio.3000186. eCollection 2019 Aug. PMID 31398186
- [Background] Poltoratski S, Tong F. Resolving the Spatial Profile of Figure Enhancement in Human V1 through Population Receptive Field Modeling. J Neurosci. 2020 Apr 15;40(16):3292-3303. doi: 10.1523/JNEUROSCI.2377-19.2020. Epub 2020 Mar 5. PMID 32139585
- [Background] Poltoratski S, Ling S, McCormack D, Tong F. Characterizing the effects of feature salience and top-down attention in the early visual system. J Neurophysiol. 2017 Jul 1;118(1):564-573. doi: 10.1152/jn.00924.2016. Epub 2017 Apr 5. PMID 28381491